CLINICAL TRIAL: NCT02033421
Title: Beta-lactam Pharmacokinetic Profiles in Patients With Infective Endocarditis
Brief Title: Beta-lactam Pharmacokinetics in Patients With Infective Endocarditis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristina Öbrink-Hansen, MD, ph.d.-student, University of Aarhus
Other Study IDs: IE-100-2014; IE-150-2014
Record Dates: First submitted 2013-12-18; First posted 2014-01-10 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis; Therapeutic drug monitoring
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacokinetics Beta-lactam antibiotics: Patients with infective endocarditis treated with Beta-lactam antibiotics

SUMMARY:
The recommended length of antibiotic treatment to patients with infective endocarditis is 4-6 weeks. All patients receive the same dosis except for those with renal impairment who receive a smaller dose. For Beta-lactam antibiotics, a plasma concentration above the minimal inhibitory concentration (MIC) for at least 50% of the time in a dosing interval maximize bactericidal activity. To estimate the time for which the antibiotic concentration is above the MIC (T>MIC) and to see if there might be a relationship between the concentration of antibiotics and possible side-effects, toxicity and treatment failure, all patients admitted with infective endocarditis will be followed and have two blood tests withdrawn once a week during antibiotic treatment, an expected average of 5 weeks.

DETAILED DESCRIPTION:
Comorbidity is common in patients admitted with infective endocarditis and this may effect the pharmacokinetics of antibiotics. The same dose of antibiotics may therefore result in different plasma concentrations in different patients, and this might influence possible side-effects, toxicity and treatment failure.

To investigate this further, all patients admitted with infective endocarditis, treated with Beta-lactam antibiotics, will be followed and have two blood tests withdrawn once a week during antibiotic treatment, an expected average of 5 weeks. Beta-lactam is administered every 6th hour. The first blood test will be withdrawn three hours after antibiotic infusion. The second blood test will be withdrawn right before the next antibiotic infusion. There is no intervention in the study, the results are observational. The results will contribute to assess the efficacy and quality of the treatment and help evaluate whether plasma concentration of antibiotics should be taken as a routine blood test every week in patients with infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with infective endocarditis
* Treatment with Beta-lactam antibiotics

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with infective endocarditis at the Department of Cardiology, Aarhus University Hospital, Denmark, treated with beta-lactam antibiotics.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Blood-plasma concentration of Beta-lactam antibiotics | Once a week during antibiotic treatment, an expected average of 5 weeks
  The first blood test will be withdrawn within a week after initiation of antibiotic therapy. The next blood test will be taken approximately 7 days after the first one and so forth once a week, until the termination of antibiotic treatment, an expected average of 5 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wiggers, Md, D.Sc, Principal Investigator — Department of cardiology, Aarhus University hospital, Denmark
Locations (1):
- Department of cardiology, Aarhus University Hospital, Aarhus N, Denmark, Denmark